CLINICAL TRIAL: NCT05214040
Title: Vitamin D Insufficiency inVestigation Among hospitaLizeD Inpatients
Acronym: VIVALDI
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 4750685
Record Dates: First submitted 2021-12-21; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Hypovitaminosis D
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypovitaminosis D is common in the adult population, it affects at least 1 billion people worldwide, and in particular 80% of the French population according to the National Institute for Public Health Surveillance. Hypovitaminosis D is accompanied or complicated by deleterious health manifestations such as bone, immune and cancer diseases, neuromuscular disorders and a propensity to fall, for example. Hypovitaminosis D has also been associated with more complicated care pathways (increase in the severity of the reason for hospitalization, length of hospitalization, risk of in-hospital death). Prevention of these clinical events depends on correcting vitamin D status.

In sick, dependent or fragile adults, natural intakes are generally insufficient. It is indeed accepted that hypovitaminosis D may not be treated effectively by dietary measures or by simple exposure to the sun in French latitudes. Drug supplementation is therefore necessary, with the objective of achieving a target concentration of circulating 25-hydroxyvitamin D (25 (OH) D) of 75 nmol / L (30 ng / mL) in this population.

Vitamin D supplementation, when properly conducted, corrects hypovitaminosis D, and has been associated with improved prognosis, especially life-saving, in therapeutic trials versus placebo. Such results lead the investigators to suggest that the identification and correction of hypovitaminosis D in hospitalized patients could represent a simple, effective and inexpensive strategy for improving hospital care pathways. In this perspective, the first step is to determine the prevalence, severity and clinical profile of hospitalized patients with hypovitaminosis D, as well as their course of care. To the investigators knowledge, there are no large-scale studies based on real-life data on this subject.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* have had a dosage of circulating 25-hydroxyvitamin D (plasma or serum) in a HUGO establishment
* consultant or hospitalized between 01/01/2015 and 12/31/2019 in one of the participating HUGOs.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients meeting the eligibility criteria over the study period.
Sampling Method: Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence and depth of hypovitaminosis D | baseline
  the prevalence of hypovitaminosis D will be calculated for each of the 3 definition thresholds for hypovitaminosis D found in the literature: ≤ 75 nmol/L, ≤ 50 nmol/L and ≤ 25 nmol/L.

SECONDARY OUTCOMES:
Clinical profile | baseline
  The clinical profile will be determine by the data provided by the physician during the hospitalization or the consultation
Length of hospitalisation | baseline
  determine whether the circulating 25-hydroxyvitamin D concentration is associated with the length of hospitalization in days
Mortality | baseline, 14 and 28 days, 3 and 6 months after the dosage
  determine whether the circulating 25-hydroxyvitamin D concentration is associated with the death occurring during hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Cédric ANNWEILER, MD,PhD, Principal Investigator — Angers University Hospital